CLINICAL TRIAL: NCT06478238
Title: A Prospective Single Arm Clinical Trial of Calcium Folinate in the Treatment of Spastic Paraplegia 56
Brief Title: Calcium Folinate Treatment of Spastic Paraplegia 56
Acronym: CFT-SPG56
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Li Cao, Head of the Department of Neurology, Shanghai 6th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-058-(1)
Record Dates: First submitted 2024-06-08; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Hereditary Spastic Paraplegia
MeSH Terms: conditions — Spastic Paraplegia, Hereditary | interventions — Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- calcium folinate treatment group (Experimental): Drug: calcium folinate Phase I: calcium folinate infusion intravenously for 5 consecutive days at a dose of 1mg/kg/day in two divided doses per day. Then it was changed to oral administration at a dose of 2mg/kg/day during hospitalization.
  Phase II: long-term oral medication at a dose of 2mg/ kg/day in two daily doses.
  Interventions: Drug: calcium folinate

INTERVENTIONS:
Drug: calcium folinate — Intravenous infusion and/or oral therapy

SUMMARY:
SPG56 is one of the complicated and early-onset HSP subtypes caused by genetic mutations in CYP2U1. So far, there is no standardized and specific clinical therapy for SPG56. The goal of this clinical trial is to explore the efficacy and safety of calcium folinate in the treatment of SPG56 patients.

This study is prospective, open-label and single arm and this trial will last for 6 years. A total of 10 patients will participate and they will receive calcium folinate treatment and professional clinical evaluation regularly.

ELIGIBILITY:
Inclusion Criteria:

1. Patients meet the clinical diagnostic standard of hereditary spastic paraplegia (HSP);
2. Spastic paraplegia type 56 (SPG56) was diagnosed by CYP2U1 pathogenic mutation;
3. Patients are willing to participate in clinical trials and able to understand and comply with the research program.

Exclusion Criteria:

1. Patients are allergic to the drugs involved in the study;
2. Other neurological diseases likely affecting the evaluation of study treatment;
3. Other medical conditions such as: heart disease, tumor, blood disease, liver disease, kidney disease, etc. in the past 1 year;
4. Pregnancy or lactating women or subjects who are unable to use appropriate contraception during the trial;
5. Participating in another study drug trial and used the investigational drug in the past 30 days;
6. Subjects have poor compliance or other factors that are not suitable for participating in the clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2030-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
GMFM-88 | At the end of the 5-year follow-up period
  The change in the Gross Motor Function Measure-88 (GMFM-88) score from baseline (range: 0-264, higher scores mean a better outcome).

SECONDARY OUTCOMES:
SPRS score | At the end of the 5-year follow-up period
  The change in the Spastic Paraplegia Rating Scale (SPRS) score from baseline (range: 0-52, higher scores mean a worse outcome).
MMSE score | At the end of the 5-year follow-up period
  The change in the Mini-Mental State Examination (MMSE) score from baseline (range: 0-30, higher scores mean a better outcome).
Laboratory indicators | At the end of the 5-year follow-up period
  The change in the Laboratory indicators (blood biochemistry, lipid metabolism, folate, etc) and the number of participants with abnormal laboratory indicators.
Cranial CT/MRI | At the end of the 5-year follow-up period
  The change in the cranial CT/MRI from baseline.
Gait examination | At the end of the 5-year follow-up period
  The change in the gait examination from baseline.
MoCA score | At the end of the 5-year follow-up period
  The change in the Montreal Cognitive Assessment (MoCA) score from baseline (range: 0-30, higher scores mean a better outcome).
High density electroencephalogram | At the end of the 5-year follow-up period
  The change in the high density electroencephalogram from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai 6th People's Hospita, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided